CLINICAL TRIAL: NCT06722456
Title: Set-up of Mass Spectrometry-based Stool Tests for Improving the Diagnosis and Management of Inflammatory Bowel Disease
Brief Title: Assessment of Non-invasive Tools for Detecting Active Inflammatory Bowel Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Jean-François Beaulieu (Other)
Responsible Party: Sponsor-Investigator, Jean-François Beaulieu, Professor, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Other Study IDs: 90-18A
Record Dates: First submitted 2024-11-28; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Disease (IBD); Crohn Disease (CD); Ulcerative Colitis (UC)
Keywords: Diagnosis; Non-invasive; Remission
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- IBD in remission: Patient affected with an inflammatory bowel disease that is considered in remission.
  Interventions: Diagnostic Test: Analysis of protein signatures in stool samples
- IBD active: Patient affected with an inflammatory bowel disease that is considered under an active state.
  Interventions: Diagnostic Test: Analysis of protein signatures in stool samples
- IBD not classified: Patient affected with an inflammatory bowel disease that is difficult to classify as active or in remission.
  Interventions: Diagnostic Test: Analysis of protein signatures in stool samples

INTERVENTIONS:
Diagnostic Test: Analysis of protein signatures in stool samples — Stool protein signatures are to be established in parallel to standard clinical evaluation of the intestinal inflammatory activity.

SUMMARY:
Part of the success of the treatment of people living with inflammatory bowel diseases (IBD) depends on the information that the doctor can obtain from the different clinical tests. Some of these tests are invasive such as the colonoscopy but other such the fecal calprotectin test, which measures intestinal inflammation, are non-invasive and useful to evaluate the success of the treatments. Unfortunately, the results from the non-invasive tests are not always clear and need to be complete with invasive tests for the right diagnosis.

The aim of this research is to test new stool markers for assisting the gastroenterologist to diagnose inflammatory bowel conditions including Crohn's disease (CD) and ulcerative colitis (UC) and to carefully monitoring the effects of medications on remission. We are using applications based on the use of mass spectrometry for identifying the proteins that are released by the host in the stools. We have identified more than 400 proteins in total. Based on informatics, we have been able to produce lists of unique stool proteins that can rapidly inform the doctor if the person has an IBD, whether it is a CD or an UC and, more importantly for the treatment, if the IBD is active or in remission.

The purpose of this study is to validate these protein markers in a blind test, where the real diagnosis will only be revealed after the analysis of the samples.

This study will bring a new power tool to assist the gastroenterologist in the treatment of people living with IBD.

ELIGIBILITY:
Inclusion Criteria:

* Be affected with one of the two main inflammatory bowel diseases (Crohn's disease of ulcerative colitis).
* Be invited to participate on the base of a routine follow up by their gastroenterologist.
* Be scheduled for a calprotectin test and a colonoscopy.
* Accept to participate and provide an extra stool sample for analysis.

Exclusion Criteria:

* Having no history of inflammatory bowel disease.
* Be affected with an history of gastrointestinal disease other than Crohn disease or ulcerative colitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed by a gastroenterologist at the CIUSS de l'Estrie-CHUS.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Scoring intestinal inflammation from stool protein analyses | From enrolment to the end of full data compilation, assessed up to 15 months
  Assessing activity in patients affected with Crohn's disease or ulcerative colitis on a 0 to 1.0 score (0 as best score for remission to 1.0 as maximal score for activity) for evaluating intestinal inflammation by proteomics analysis of stools relative to standard clinical criteria (symptoms and results from colonoscopy, histopathology and fecal calprotectin).

SECONDARY OUTCOMES:
To compare activity scores deduced from proteomics analyses to the results from colonoscopy and pathology. | From enrolment to the end of full data compilation, assessed up to 15 months
  Assessing activity in patients affected with Crohn's disease or ulcerative colitis on a 0 to 1.0 score for evaluating intestinal inflammation by proteomics analysis of stools relative to the results from colonoscopy and histopathology.
To compare activity scores deduced from proteomics analyses to the results from pathology. | From enrolment to the end of full data compilation, assessed up to 15 months
  Assessing activity in patients affected with Crohn's disease or ulcerative colitis on a 0 to 1.0 score for evaluating intestinal inflammation by proteomics analysis of stools relative to the results from histopathology.
To compare activity scores deduced from proteomics analyses to the results from fecal calprotectin. | From enrolment to the end of full data compilation, assessed up to 15 months
  Assessing activity in patients affected with Crohn's disease or ulcerative colitis on a 0 to 1.0 score for evaluating intestinal inflammation by proteomics analysis of stools relative to the results of fecal calprotectin.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche of the CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlies results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication
Access Criteria: Study protocol and SAP will be accessible from the publication.

REFERENCES:
- [Background] Shajari E, Gagne D, Malick M, Roy P, Noel JF, Gagnon H, Brunet MA, Delisle M, Boisvert FM, Beaulieu JF. Application of SWATH Mass Spectrometry and Machine Learning in the Diagnosis of Inflammatory Bowel Disease Based on the Stool Proteome. Biomedicines. 2024 Feb 1;12(2):333. doi: 10.3390/biomedicines12020333. PMID 38397935
- See also: Laboratory webpage on research pertaining to inflammatory bowel disease. — https://labppi.wordpress.com/inflammatory-bowel-diseases/